CLINICAL TRIAL: NCT03600675
Title: Determinants of Bone Mineral Density and Metabolic Syndrome in South Asian Indian Men
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Other Study IDs: 1604004460R001
Record Dates: First submitted 2018-03-14; First posted 2018-07-26 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
Keywords: Body composition; Abdominal fat; Inflammatory cytokines; Bone markers; Bone mineral density
MeSH Terms: conditions — Osteoporosis | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- South Asian Indians: No intervention will be applied for any group
  Interventions: Other: No intervention element, observational study.
- Caucasians: No intervention will be applied for any group
  Interventions: Other: No intervention element, observational study.

INTERVENTIONS:
Other: No intervention element, observational study. — No intervention will be applied to any group. It is an observational study and all measurements are collected during one visit.
  Other Names: Observational Study

SUMMARY:
This study aims to examine the association between body composition with bone density and risk factors for cardiovascular disease and type 2 diabetes. South Asian Indians have a lower bone density and a higher likelihood to develop metabolic syndrome (MetS) compared to Caucasians. MetS is a cluster of metabolic abnormalities that predispose an individual to cardiovascular disease and type 2 diabetes. This study will understand if the metabolic and biochemical markers ( Indicators of bone building and breaking in the blood and urine, Lipids and other proteins) explain both low BMD and MetS in SAI men

DETAILED DESCRIPTION:
There is a rising minority population in the United States and South Asians make up the largest growing sub population. Health concerns in the minority population are several of which metabolic syndrome (MetS) and low bone mineral density (BMD) are important. Interestingly research in the past decade is beginning to suggest an interplay between bone and energy metabolism. Hormones, bone proteins and cytokines that play an important role in bone metabolism are also altered in metabolic syndrome, suggesting that both these

conditions may share a common etiology. Hence the primary question in this study would be to assess whether bone is altered in the South Asian population in the United States and whether hormones or other proteins regulating bone influence metabolic syndrome outcomes in the South Asians, specifically the South Asian Indian population. There is also an altered body composition in the South Asian Indian population with a greater visceral adiposity. Greater visceral adipose tissue (VAT) is associated in both the pathogenesis of metabolic syndrome and low BMD, possibly due to release of pro inflammatory cytokines. Interestingly several factors that are involved in the etiology of low BMD such as a greater visceral adiposity, high serum pro inflammatory cytokines, altered hormonal milieu such as low 25 hydroxy vitamin D (25OHD) and high parathyroid hormone (PTH), low osteocalcin levels, low calcium and high carbohydrate diet may share a relationship with MetS outcomes. The South Asian population has all the above-mentioned biochemical and metabolic alterations and it would be interesting to examine this in an immigrant Asian population residing in the USA. The investigators propose to examine 30 South Asian Indians between the ages of 30-50 years, using 30 resident Caucasian men as controls. Bone measures such as BMD and bone mineral content will be measured at radius, trochanter, hip and tibia and body composition including lean mass, fat mass, android fat and gynoid fat will be assessed using the Dual X ray energy absorptiometry (DXA). Biochemical measures including a complete metabolic panel, PTH, 25OHD, osteocalcin and other bone markers, and pro inflammatory cytokines will be measured in the serum. Investigators hypothesize that South Asian Indian men will have a lower BMD and higher MetS risk factors compared to age and BMI matched Caucasian men. Investigators further propose that common biochemical and metabolic alterations will underlie both low BMD and MetS outcomes in SAI population, but not in the Caucasian population. Identification of common determinants will help design a single future interventional trial that will target both MetS and bone health in the SA population

Specific Aim 1 To determine whether Bone Mineral Density (BMD) at weight-bearing and non weight-bearing sites is lower in age- and weight-matched SAI compared to white men.

It is hypothesized that SAI men will have lower BMD at weight-bearing sites compared to age and BMI-matched white men.

Specific Aim 2 To determine whether body composition influences Bone Mineral Density in SAI men.

It is hypothesized that greater abdominal adiposity, specifically visceral fat, influences BMD in SAI men compared to age- and BMI-matched white men.

Specific Aim 3 To examine the hormonal, inflammatory, and dietary determinants of Bone Mineral Density and MetS in SAI compared to white men.

It is hypothesized that the hormonal, inflammatory, and dietary determinants of both MetS and low BMD will be similar in the SAI men but not in the white men.

This study will involve one single visit. The following will be conducted during this visit:

* This visit will last for about 2 hours
* Blood draw- Four 5 ml tubes of blood will be collected via venipuncture
* Spot urine sample collection
* Measurement of height, weight, blood pressure, waist circumference
* Completion of study questionnaires
* DXA scan

ELIGIBILITY:
Inclusion Criteria:

* South Asian Indian and Caucasian males
* 20 and 50 years of age
* BMI range 23 - 35 kg/m2

Exclusion Criteria:

* An individual is unwilling to sign the informed consent document.
* A physician states that a participant is not able to participate in the study.
* Individuals with the presence of any acute illness in the past month.
* Individuals with preexisting chronic medical conditions such as diabetes (type I and II), cancer, other metabolic disorders.
* Individuals who are using medications known to influence bone, blood glucose, lipids,and blood pressure.
* Individuals who had a history of major diseases, such as cardiac, diabetes, renal, or evidence of cancer, in the past year.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: South Asians Indians are defined as those who can trace their ancestry to Bangladesh, Bhutan, India, the Maldives, Nepal, Pakistan, and Sri Lanka.
  Caucasians are defined as non-Hispanic who do not belong to any other ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density ( g/cm2) | 1 day at baseline
  Baseline differences in BMD in 2 groups
Total Body fat ( kg) | 1 day at baseline
  Using the total body scan from the DXA , fat mass will be assessed
Lean mass ( Kg) | 1 day at baseline
  Using the total body scan from the DXA , lean mass will be assessed
Visceral adipose tissue - VAT ( kg) | 1 day at baseline
  Using the total body scan from the DXA ,VAT mass will be assessed

SECONDARY OUTCOMES:
Interleukin-6 ( IL-6)- pg/mL | 1 day at baseline
  Serum levels will be assayed
Monocyte Chemoattractant protein-1 ( MCP-1)- ng//mL | 1 day at baseline
  Serum levels will be assayed
C- Reactive Protein ( CRP)-mg/L | 1 day at baseline
  Serum levels will be assayed
Adiponectin- ng/mL | 1 day at baseline
  Serum levels will be assayed
Lipid profile | 1 day
  Serum levels of HDL, LDL, Total cholesterol and triglycerides will be assayed ( mg/dL)
Blood pressure | 1 day
beta-C-terminal telopeptide (CTx) - ug/L | 1 day
  Serum levels will be assayed
Parathyroid hormone- pg/mL | 1 day
  Serum levels will be assayed
25 hydroxy vitamin D- ng/ML | 1 day
  Serum levels will be assayed
Osteocalcin ( total)- ng/mL | 1 day
  Serum levels will be assayed

CONTACTS AND LOCATIONS:
Overall Officials: Deeptha Sukumar, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University Nutrition Sciences Research Lab, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided